CLINICAL TRIAL: NCT01600092
Title: A Double-blind, Randomized, Controlled, Multicenter Study to Evaluate the Safety, Tolerability, and Immunogenicity of a New Formulation of RotaTeq™
Brief Title: A Study of the Immunogenicity, Tolerability, and Safety of a New Formulation of RotaTeq™ in Infants (V260-035)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: V260-035
Record Dates: First submitted 2012-05-14; First posted 2012-05-16 (Estimated); Results first posted 2015-03-19 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-10

CONDITIONS: Rotavirus Gastroenteritis
MeSH Terms: interventions — Rotavirus Vaccines

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- RotaTeq™ Experimental Formulation (Experimental): Three 2.0 mL oral doses of RotaTeq™ experimental formulation. Vaccination 1 will be administered between 6 and 12 weeks of age and the third vaccination will be administered before 32 weeks of age. Each vaccination will be separated from the next by ≥ 4 weeks (28 days)
  Interventions: Biological: RotaTeq™ experimental formulation
- RotaTeq™ Existing Formulation (Active Comparator): Three 2.0 mL oral doses of RotaTeq™ existing formulation. Vaccination 1 will be administered between 6 and 12 weeks of age and the third vaccination will be administered before 32 weeks of age. Each vaccination will be separated from the next by ≥ 4 weeks (28 days).
  Interventions: Biological: RotaTeq™ existing formulation

INTERVENTIONS:
Biological: RotaTeq™ experimental formulation
  Other Names: V260
  Arms: RotaTeq™ Experimental Formulation
Biological: RotaTeq™ existing formulation
  Other Names: V260
  Arms: RotaTeq™ Existing Formulation

SUMMARY:
A study to compare safety, tolerability, and immunogenicity of a new formulation of RotaTeq™ with the existing formulation in infants. The primary hypothesis of the study is that the new formulation will be noninferior to the existing formulation on the basis of immunogenicity.

ELIGIBILITY:
Inclusion Criteria:

* Parent or legal guardian agrees to have infant participate by giving written informed consent

Exclusion Criteria:

* History of congenital abdominal disorders, prior rotavirus gastroenteritis, chronic diarrhea, failure to thrive, or abdominal surgery
* History of intussusception
* Known or suspected impairment of immunological function, including Severe

Combined Immunodeficiency (SCID)

* Prior administration of any rotavirus vaccine
* Clinical evidence of active gastrointestinal illness, with the exception of well-controlled gastroesophageal reflux disease (GERD)
* Receipt of 1) systemic corticosteroids (≥ 2mg/kg total daily dose of prednisone or equivalent) for 14 consecutive days or more since birth, or 2) systemic corticosteroids ≥ 2mg/kg/dose within 7 days prior to the administration of the first dose of study vaccine. Participant using non-systemic corticosteroids will be eligible for vaccination.
* Residing in a household with an immunocompromised person
* Prior receipt of a blood transfusion or blood products, including immunoglobulins
* Participation in another interventional study within 14 days prior to the first study vaccination or expected anytime during the study
* Receipt of investigational inactivated vaccines within 14 days or investigational live vaccines within 28 days prior to the first study vaccination or expected anytime during the study

Ages: 6 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1020 (Actual)
Dates: Start 2013-04-29 (Actual); Primary Completion 2014-03-25 (Actual); Study Completion 2014-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Martinon-Torres F, Greenberg D, Varman M, Killar JA, Hille D, Strable EL, Stek JE, Kaplan SS. Safety, Tolerability and Immunogenicity of Pentavalent Rotavirus Vaccine Manufactured by a Modified Process. Pediatr Infect Dis J. 2017 Apr;36(4):417-422. doi: 10.1097/INF.0000000000001511. PMID 28141698
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=V260-035&kw=V260-035&tab=access

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 1039 participants were screened
Period: Overall Study
Arm/Group | RotaTeq™ Experimental Formulation | RotaTeq™ Existing Formulation
Started | 513 | 507
Received at Least 1 Vaccination | 510 (1 participant received RotaTeq™ existing formulation as their first vaccination) | 504
Received All 3 Vaccinations | 500 | 494
Completed | 495 | 491
Not Completed | 18 | 16
Not completed — Adverse Event | 2 | 0
Not completed — Lost to Follow-up | 4 | 6
Not completed — Withdrawal by parent/guardian | 8 | 6
Not completed — Physician Decision | 1 | 1
Not completed — Randomized but not vaccinated | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RotaTeq™ Experimental Formulation | RotaTeq™ Existing Formulation | Total
Number analyzed (Participants) | 513 | 507 | 1020
Age, Continuous [Mean (Standard Deviation); unit: Weeks] | 8.4 (1.4) | 8.3 (1.4) | 8.3 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 232 | 240 | 472
  Male | 281 | 267 | 548

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titer of Serum Neutralizing Antibody Response to Human Rotavirus Serotypes G1, G2, G3, G4, and P1A[8]
Time Frame: 42 days after vaccination 3 (up to 185 days)
Population: Participants who received the 3 scheduled doses of study vaccine, did not have important protocol deviations, and had follow-up results for the endpoint
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | RotaTeq™ Experimental Formulation | RotaTeq™ Existing Formulation
Number analyzed (Participants) | 480 | 482
Titer
  Serotype G1 | 99.8 [89.7 to 111.1] | 106.1 [94.6 to 119.0]
  Serotype G2 | 30.0 [27.0 to 33.3] | 26.3 [23.7 to 29.1]
  Serotype G3 | 82.8 [74.2 to 92.5] | 25.2 [22.6 to 28.1]
  Serotype G4 | 78.9 [72.3 to 86.1] | 71.5 [65.4 to 78.1]
  Serotype P1A[8] | 106.9 [96.5 to 118.4] | 90.1 [80.2 to 101.2]
Statistical Analysis 1: Comparison: RotaTeq™ Experimental Formulation vs RotaTeq™ Existing Formulation; Serotype G1; Test type: Non-Inferiority or Equivalence — Non-inferiority required that the lower bound of the 2-sided 95% confidence interval of the GMT ratio is >0.67; GMT Ratio (Experimental/Existing) = 0.92, 95% CI 2-sided [0.79 to 1.07] — GMTs and GMT ratio were based on a model with terms for treatment and country, with the constraint that the mean baseline value is the same for both treatment groups
Statistical Analysis 2: Comparison: RotaTeq™ Experimental Formulation vs RotaTeq™ Existing Formulation; Serotype G2; Test type: Non-Inferiority or Equivalence — Non-inferiority required that the lower bound of the 2-sided 95% confidence interval of the GMT ratio is >0.67; GMT Ratio (Experimental/Existing) = 1.15, 95% CI 2-sided [0.99 to 1.33] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: RotaTeq™ Experimental Formulation vs RotaTeq™ Existing Formulation; Serotype G3; Test type: Non-Inferiority or Equivalence — Non-inferiority required that the lower bound of the 2-sided 95% confidence interval of the GMT ratio is >0.67; GMT Ratio (Experimental/Existing) = 3.20, 95% CI 2-sided [2.75 to 3.74] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: RotaTeq™ Experimental Formulation vs RotaTeq™ Existing Formulation; Serotype G4; Test type: Non-Inferiority or Equivalence — Non-inferiority required that the lower bound of the 2-sided 95% confidence interval of the GMT ratio is >0.67; GMT Ratio (Experimental/Existing) = 1.06, 95% CI 2-sided [0.94 to 1.20] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: RotaTeq™ Experimental Formulation vs RotaTeq™ Existing Formulation; Serotype P1A[8]; Test type: Non-Inferiority or Equivalence — Non-inferiority required that the lower bound of the 2-sided 95% confidence interval of the GMT ratio is >0.67; GMT Ratio (Experimental/Existing) = 1.16, 95% CI 2-sided [1.00 to 1.35] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Number of Participants With Tier-1 Adverse Events: Diarrhea, Vomiting, Elevated Temperature, and Irritability
Description: An adverse event is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study vaccine, whether or not considered related to the use of the product. Any worsening of a preexisting condition which is temporally associated with the use of the study vaccine is also an adverse event. Protocol-defined Tier-1 adverse events to be collected up to 7 days after any vaccination were diarrhea, vomiting, elevated temperature (rectal >=38.1° C, >=100.5° F), and irritability.
Time Frame: Up to 7 days after any vaccination (up to 147 days)
Population: Participants who received at least one dose of study vaccine. Participants were assigned to treatment groups based on the vaccine received as the first dose.
Measure: Number; unit: Participants
Arm/Group | RotaTeq™ Experimental Formulation | RotaTeq™ Existing Formulation
Number analyzed (Participants) | 509 | 505
Participants
  Diarrhea | 144 | 128
  Vomiting | 84 | 92
  Elevated temperature | 217 | 223
  Irritability | 58 | 64

3. Secondary Outcome: Number of Participants With Tier-1 Adverse Events: Intussusception
Description: The protocol-defined Tier-1 adverse event to be collected for the duration of the study (up to Day 185) was intussusception
Time Frame: Up to Day 185
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | RotaTeq™ Experimental Formulation | RotaTeq™ Existing Formulation
Number analyzed (Participants) | 509 | 505
Participants | 2 | 0

4. Secondary Outcome: Geometric Mean Titer of Serum Anti-Rotavirus Immunoglobulin A
Time Frame: 42 days after vaccination 3 (up to 185 days)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | RotaTeq™ Experimental Formulation | RotaTeq™ Existing Formulation
Number analyzed (Participants) | 474 | 474
Titer | 240.5 [210.4 to 274.8] | 235.5 [204.1 to 271.8]

5. Secondary Outcome: Percentage of Participants With >=3-fold Rise From Baseline in GMT of Serum Neutralizing Antibody to Human Rotavirus Serotypes G1, G2, G3, G4, and P1A[8]
Time Frame: Baseline and 42 days after vaccination 3 (up to 185 days)
Population: Participants who received the 3 scheduled doses of study vaccine, did not have important protocol deviations, and had baseline and follow-up results for the endpoint
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | RotaTeq™ Experimental Formulation | RotaTeq™ Existing Formulation
Number analyzed (Participants) | 480 | 481
Percentage of participants
  Serotype G1 | 56.0 [51.5 to 60.5] | 53.8 [49.3 to 58.4]
  Serotype G2 | 30.4 [26.3 to 34.7] | 26.8 [22.9 to 31.0]
  Serotype G3 | 65.8 [61.4 to 70.1] | 33.3 [29.1 to 37.7]
  Serotype G4 | 58.3 [53.8 to 62.8] | 49.7 [45.1 to 54.3]
  Serotype P1A[8] | 49.6 [45.0 to 54.2] | 42.6 [38.2 to 47.2]

ADVERSE EVENTS:
Time Frame: All adverse events: up to 42 days after any vaccination; serious adverse events, deaths, and intussusception: up to Day 185
Description: The participants at risk includes participants who received at least one dose of study vaccine and had follow-up
Arm/Group | RotaTeq™ Experimental Formulation | RotaTeq™ Existing Formulation
Serious Adverse Events (participants affected / at risk) | 20/508 | 12/499
Other Adverse Events (participants affected / at risk) | 398/508 | 385/499
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RotaTeq™ Experimental Formulation (N=508) | RotaTeq™ Existing Formulation (N=499)
Intussusception (Gastrointestinal disorders) | 2 (2) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 1 (1) | 1 (1)
Bronchiolitis (Infections and infestations) | 3 (3) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0)
Parainfluenzae virus infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypersomnia (Nervous system disorders) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RotaTeq™ Experimental Formulation (N=508) | RotaTeq™ Existing Formulation (N=499)
Constipation (Gastrointestinal disorders) | 30 (33) | 22 (29)
Diarrhoea (Gastrointestinal disorders) | 173 (307) | 156 (276)
Vomiting (Gastrointestinal disorders) | 102 (175) | 107 (180)
Pyrexia (General disorders) | 151 (211) | 152 (231)
Conjunctivitis (Infections and infestations) | 27 (35) | 25 (25)
Nasopharyngitis (Infections and infestations) | 79 (106) | 83 (113)
Otitis media (Infections and infestations) | 20 (26) | 29 (33)
Rhinitis (Infections and infestations) | 42 (53) | 40 (56)
Upper respiratory tract infection (Infections and infestations) | 78 (97) | 67 (87)
Irritability (Psychiatric disorders) | 65 (98) | 77 (113)
Cough (Respiratory, thoracic and mediastinal disorders) | 36 (39) | 44 (50)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation.